CLINICAL TRIAL: NCT01401946
Title: Soy Isoflavone Tablets: Effects on Questionnaire and Actigraphic Measures of Sleep, Symptoms as Measured by the Women's Health Questionnaire and Cognitive Function as Measured by Computerized Cognitive Performance Tests in Menopausal Women
Brief Title: Soy Isoflavone Tablets: Effects on Sleep, Quality of Life, Symptoms and Cognitive Function in Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Quentin R. Regestein, Brigham & Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99-004-P
Record Dates: First submitted 2010-12-08; First posted 2011-07-26 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- soy isoflavones (Active Comparator)
  Interventions: Drug: soy isoflavones
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: soy isoflavones
  Arms: soy isoflavones
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study was done to elucidate relationships between midlife women's self-reported hot flashes, neuropsychological symptoms, cognitive performance or sleep.

ELIGIBILITY:
Inclusion criteria:

* At least 5 hot flash episodes and/or night sweats per 24 hours

Exclusion Criteria:

* Body mass index (BMI) more than 34 kg/m2
* Hypertension
* Shift work
* Psychiatric or medical conditions that would affect outcome measures
* More than 4 caffeine drinks per day
* More than 10 cigarettes per day
* More than than 7 alcohol drinks per week

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2000-05; Primary Completion 2000-10 (Actual); Study Completion 2001-01 (Actual)

PRIMARY OUTCOMES:
Soy Isoflavone: Effects on Sleep, Symptoms, Quality of Life and Cognitive Function in Menopausal Women | Nine weeks
  Hot flashes recorded by means of 5 global estimation and daily diary measures of hot flashes and night sweats.
Soy Isoflavone: Effects on Sleep, Symptoms, Quality of Life and Cognitive Function in Menopausal Women | 9 weeks
  Symptoms recorded on the Women's Health Questionniare at baseline and 4 subsequent occasions
Soy Isoflavone Tablets: Effects on Sleep, Quality of Life, Symptoms and Cognitive Function in Menopausal Women | 9 weeks
  Subjective sleep measured by average questionnaire item scores recorded each morning for a week, repeated at baseline and 4 subsequent times
Soy Isoflavone Tablets: Effects on Sleep, Quality of Life, Symptoms and Cognitive Function in Menopausal Women | 9 weeks
  Cognitive function measured by computerized cognitive performance tests of motor speed, switching attention, continuous performance and Stroop color-word tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States